CLINICAL TRIAL: NCT05134129
Title: Correlation Between Targeted Hemoglobin A1C Levels and Prevention of Recurrent Cardiovascular Events in Type 2 Diabetes After Coronary Intervention
Brief Title: Correlation Between Targeted HbA1c Values and Prevention of Recurrent Cardiovascular Events in Type 2 Diabetes After PCI
Acronym: CATHEDRAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Other Study IDs: CATHEDRAL
Record Dates: First submitted 2021-08-10; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus; Percutaneous Coronary Intervention
Keywords: Glycated Hemoglobin; Percutaneous Coronary Intervention; Metabolomics; Diabetes Mellitus; Cardiovascular Risk
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples were taken for metabolomics study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes is a leading social and economic burden in the world. It is the main reason of macrovascular disease incidence and mortality. Prospective studies have demonstrated that high glycosylated hemoglobin (HbA1C) levels are associated with an increased risk of cardiovascular events in a population of diabetic patients without a history of coronary artery disease. Further, the predictive value of high preprocedural glycemia levels has been reported in diabetic patients undergoing percutaneous coronary intervention (PCI). The aim of the present study was to assess the predictive value of preprocedural HbA1C levels for cardiovascular complications in a large population of diabetic patients undergoing PCI with stent implantation. Glycosylated hemoglobin (HbA1c) reflects the average blood sugar level in the past 2-3 months. As glycosylated hemoglobin has been clinically tested and standardized internationally, increasing evidence is recommended for routine monitoring in diabetes care. The American Diabetes Association (ADA) suggested that in the treatment of diabetes, blood sugar control should control HbA1c level below 6.5%. Although，there is evidence that controlling blood glucose can reduce the incidence of microvascular complications, in the past three trials, intensive glycemic control did not significantly reduce adverse CV events in patients with onger duration of diabetes.Therefore, most primary and secondary prevention guidelines recommend HbA1c below 6.5% or 7% to prevent adverse cardiovascular outcomes in patients with diabetes mellitus. The optimal target level of glycosylated hemoglobin is still hotly debated. In addition, there is still lack of evidence for the level of HbA1c in patients with major vascular disease history in secondary prevention of recurrence cardiovascular events.

Therefore, to explore and determine the optimal level of blood glucose control is the focus of controversy in preventing recurrence cardiovascular events in diabetic patients. Investigator will combine epidemiology and metabolomics to study the effect of glycosylated hemoglobin on secondary cardiovascular events, and further determine whether to strengthen hypoglycemic treatment after PCI.

DETAILED DESCRIPTION:
This is a longitudinal cohort study including retrospective study, prospective study and nested case-control study.The first cross-sectional survey was conducted in 2021.

ELIGIBILITY:
Inclusion Criteria:

- 1. Age ≥ 18, male or female;

2. all patients with diabetes combined with PCI operation;

Exclusion Criteria:

* 1. Less than 18 years old

  2. Pregnancy

  3. Patients with preoperative glycosylated hemoglobin index deficiency

  4. Chronic maintenance hemodialysis patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Demographic data, cardiovascular examinations and laboratory parameters were collected from 1500 hospitalized diabetic patients with PCI. Patients younger than 18 years old, pregnant, preoperative HbA1c deletion and chronic maintenance hemodialysis were excluded. According to ADA and AHA guidelines and predetermined glycosylated hemoglobin values, based on clinical relevance, especially glycosylated hemoglobin < 6.5%, 6.5% ≤ glycosylated hemoglobin ≤ 7.0%, glycosylated hemoglobin > 7.0%, and statistical end events including patients with more than or equal to two PCI enents, patients with all-cause motality and cardiac motality.Through prospective cohort study and nested case-control study,analysis related risk factors and metabolomics molecular differences between revascularization patients and non-revascularization patients.The instrument platforms of gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS) are used to metabonomic analysis.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-04-25 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Coronary revascularization | 3 years
  Coronary revascularization includes percutaneous coronary intervention, or/and percutaneous coronary artery dilatation, or/and percutaneous coronary artery bypass grafting.
All cause mortality | 3 years
  which refers to the total death caused by various causes in a certain period.
Cardiac mortality | 3 years
  Cardiac death refers to the death caused by serious cardiac dysfunction or failure caused by heart disease or injury in a certain period.
Differential polar compound | 3 years
  Metabonomic analysis uses non targeted detection methods to detect polar compounds in blood. The characteristic peaks of detectable substances were detected by chromatographic Series platform, and then these characteristic peaks were compared with the standard library containing more than 8000 metabolites, annotated the compounds, and screened out the different metabolites between groups.
Differential lipid compounds | 3 years
  Metabonomic analysis uses non targeted detection methods to detect lipid compounds in blood. The characteristic peaks of detectable substances were detected by chromatographic Series platform, and then these characteristic peaks were compared with the standard library containing more than 8000 metabolites, annotated the compounds, and screened out the different metabolites between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Cang, MD, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital; Zheng Liu, pHD, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital; Zhicai Wang, MD, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital
Locations (1):
- Department of Cardiology,Shanghai Tenth People's Hospital, Shanghai, China